CLINICAL TRIAL: NCT05091086
Title: The Optimal Long Term Treatment Strategy of Anti-resorptive Medications
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital Yunlin Branch, Orthopedic department, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202107164MINC
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis; Bone Mineral Density
Keywords: Osteoporosis; denosumab; zoledronic acid
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: Two parallel group would be selected. One group of participants keep their denosumab treatment for 7 years. Another group of participants accept two cycles of treatment (one year of zoledronate and two years of denosumab) and complete with one year of zoledronate.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Persistent treatment of Denosumab: (Active Comparator): persistent denosumab for 7 years
  Interventions: Drug: Continuous Denosumab
- Alternating treatment of Denosumab and Zoledronic acid (Experimental): Alternating treatment with denosumab and zoledronic acid over a 7-year period: after entering the trial, patients received one year of zoledronic acid, followed by two years of denosumab, then switched back to zoledronic acid for one year, followed by another two years of denosumab, and finally received one more year of zoledronic acid.
  Interventions: Drug: Administer zoledronate and denosumab on an alternating schedule

INTERVENTIONS:
Drug: Continuous Denosumab — Active comparator: persistent treatment of denosumab.
  Arms: Persistent treatment of Denosumab:
Drug: Administer zoledronate and denosumab on an alternating schedule — In the experimental group, zoledronic acid was administered for one year, followed by two years of denosumab. This cycle was repeated, with the regimen concluding with one year of zoledronic acid.
  Arms: Alternating treatment of Denosumab and Zoledronic acid

SUMMARY:
This study is to investigate whether the alternating use of Prolia (Denosumab) and Aclasta (Zoledronic acid) can continue to increase bone density.

DETAILED DESCRIPTION:
This study intends to use a randomized trial to test whether the long-term treatment of Denosumab and Zoledronic acid can achieve sustained bone density progress and avoid the risk of rapid bone loss after the withdrawal of Denosumab.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women or men over 50 years old with osteoporosis or osteopenia leading to fractures.
2. Denosumab treatment for at least two years and less than three years (up to maximum of five doses).

Exclusion Criteria:

1. Secondary osteoporosis.
2. Metabolic bone diseases.
3. Malignancy.
4. Continuous steroid treatment, hormone therapy or other medical treatment affecting bone metabolism.
5. Patients had ever used antiosteoporosis medications other than Dmab
6. Estimated glomerular filtration rate < 35 mL/min.
7. Allergy to Zoledronate.
8. Any other contraindications to Zoledronate use.
9. History of diagnosed hypocalcemia.
10. Age greater than 80 years.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in lumbar spine bone mineral density | From enrollment to the end of treatment at 3 years

SECONDARY OUTCOMES:
Change in total hip bone mineral density | From enrollment to the end of treatment at 3 years and 7 years
Change in femoral neck bone mineral density | From enrollment to the end of treatment at 3 years and 7 years
Change in lumbar spine bone mineral density | From enrollment to the end of treatment at 7 years
Change in C-terminal telopeptide of type 1 collagen | From enrollment to the end of treatment at 3 years and 7 years
Change in Procollagen type 1 N-terminal propeptide | From enrollment to the end of treatment at 3 years and 7 years
Fractures | 3 & 7 years
  Number of Participants with clinical fractures and radiographic vertebral fractures
Change in quality of life | From enrollment to the end of treatment at 3 years and 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Yunlin branch, Douliu, Yunlin county, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
After application